CLINICAL TRIAL: NCT00139308
Title: Pilot Study of Internal Globus Pallidus or Median Centre of the Thalamus High Frequency Stimulation for the Treatment of Patients With Severe Tourette's Syndrome
Brief Title: High Frequency Stimulation of the GPi or Thalamus in Tourette's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RBM0008
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2005-08-31 (Estimated); Status verified 2005-08

CONDITIONS: Tourette's Syndrome
Keywords: Tourette's syndrome; High frequency stimulation; Globus pallidus; Thalamus
MeSH Terms: conditions — Tourette Syndrome

INTERVENTIONS:
Device: high frequency stimulation

SUMMARY:
Tourette's syndrome is a disabling neuropsychiatric disorder with major psychosocial consequences in some patients. The pathophysiology is still unknown. Some data suggest an dysfunction of limbic circuits in basal ganglia. The aim of this study is to evaluate the effect of high frequency stimulation of the internal part of the globus pallidus and/or parafascicular-median centre of the thalamus, two structures implicated in the limbic circuit, in patients with severe Tourette's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Tourette's syndrome (DSM IV)
* inducing a disability in the social and personal life
* No improvement with medical treatment
* Severe self suffering

Exclusion Criteria:

* Cognitive impairment (MMS < 24)
* Depression

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Severity of tics

CONTACTS AND LOCATIONS:
Overall Officials: Yves Agid, MD, PhD, Study Director — CIC-Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France

REFERENCES:
- [Derived] Welter ML, Mallet L, Houeto JL, Karachi C, Czernecki V, Cornu P, Navarro S, Pidoux B, Dormont D, Bardinet E, Yelnik J, Damier P, Agid Y. Internal pallidal and thalamic stimulation in patients with Tourette syndrome. Arch Neurol. 2008 Jul;65(7):952-7. doi: 10.1001/archneur.65.7.952. PMID 18625864